CLINICAL TRIAL: NCT03247465
Title: Value of Fusion of 3D Images With 2D Images, Associated With Calcification Raising During Trans Aortic Valve Implantation Procedures
Brief Title: Image Fusion and Calcification Raising in Trans Aortic Valve Implantation
Acronym: TAVI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The deadlines of the ethics committee being very long, the investigator finally wished not to carry out the project.
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC17_0114
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Symptomatic Aortic Stenosis

STUDY DESIGN:
Intervention Model Description: The 20 first included patients will be control group, the 20 following patients will be the fusion group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group "Fusion" (Experimental): Trans aortic valve replacement with usual procedure with the addition of computed tomography 3D images and calcification raising to the usual fluoroscopy images.
  Interventions: Other: Image Fusion
- Group "Control" (No Intervention): Trans aortic valve replacement with usual procedure

INTERVENTIONS:
Other: Image Fusion — Addition of computed tomography 3D images and calcification raising to the usual fluoroscopy images.
  Arms: Group "Fusion"

SUMMARY:
Aortic stenosis is one of the most common cardiology diseases. Trans aortic valve implantation (TAVI) has been developed since 2002, first to treat rejected patients from conventional surgery, then to treat high surgical risk patients and nowadays probably intermediate surgical risk patient. TAVI related complications are still recurrent and the investigators are searching a way to decrease them.

One of them could be image fusion, since it may decrease radiation exposure and contrast agent use. It may also improve valve placement position leading to decreased complications.

40 prospective and consecutive patients will be included. Participants will be divided into two groups: the 20 first included will be control group, the 20 following patients will be the fusion group. For control group TAVI procedure will be the usual one, for fusion group the procedure will be the usual one with addition of computed tomography 3D images fusion with fluoroscopy 2D images.

Main evaluation criteria will be radiation exposure, measured by dose area product (DAP). Secondary evaluation criterion will be procedural as contrast agent volume used, procedure duration, subjective usefulness of image fusion or procedure failure evaluated immediately after procedure. The investigators will also evaluated procedure induced complications as de novo pacemaker implantation, de novo left bundle branch, vascular complication, major bleeding, acute kidney failure, significant aortic regurgitation. These complications occurrence will be evaluated after 1 month follow up, during the usual following consultation.

DETAILED DESCRIPTION:
Aortic stenosis is one of the most common cardiology diseases. If untreated, symptomatic aortic stenosis rapidly leads to death. Most of the time, this disease affects old fragile people for whom conventional surgery is countered or very risky. That is why Trans aortic valve implantation has been developed since 2002, first to treat rejected patients from conventional surgery, then to treat high surgical risk patients and nowadays probably intermediate surgical risk patient. Indeed, thanks to prodigious technical and human progress, procedure induced complication have clearly decreased. But TAVI related complications are still recurrent and the investigators are searching a way to decrease them.

One of them could be image fusion, since it may decrease radiation exposure and contrast agent use correlated to acute kidney failure. It may also improve valve placement position, and the investigators know that many rhythmic (atrio-ventricular block) and valvular (significant aortic regurgitation) complications are partially due to placement mistakes. So the investigators hope that image fusion will decrease these complications.

The investigators will include 40 prospective and consecutive patients. Inclusion criterion will be all major patients admitted in Nantes CHU for transfemoral aortic valve replacement with SAPIEN® 3 valve. Exclusion criterion will be women of childbearing age without contraception, impossible written consent, judiciary protected people. After inclusion, patients will be divided into two groups: the 20 first included will be control group, the 20 following patients will be the fusion group. For control group TAVI procedure will be the usual one, for fusion group the procedure will be the usual one with addition of computed tomography 3D images fusion with fluoroscopy 2D images. The only difference during all patient medical care will be the addition of image fusion in fusion group. Before and after procedure, both groups will have the usual medical monitoring and the appropriated medical interventions to participants case.

Main evaluation criterion will be radiation exposure, measured by dose area product (DAP).

Secondary evaluation criterion will be procedural as:

* contrast agent volume used (mL),
* procedure duration (min),
* subjective usefulness of image fusion evaluated on a 0 to 3 scale
* procedure failure : death, more than one valve implantation, valve dysfunction (mean trans-valvular gradient > 20 mmHg or moderate to severe aortic regurgitation) These criterions will be evaluated immediately after procedure.

The investigators will also evaluated procedure induced complications as:

* de novo pacemaker implantation
* de novo left bundle branch
* non minor vascular complication on VARC-2 definition
* major bleeding (BARC 3 or 5)
* acute kidney failure (AKIN 2 or 3)
* significant aortic regurgitation ≥ 2/4 These complications occurrence will be evaluated after 1 month follow up, during the usual following consultation with echocardiography.

Then differences between will be tested with appropriated statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in Nantes CHU for trans fermoral aortic valve replacement with SAPIEN 3® device
* Patient who accepted to participate to the study

Exclusion Criteria:

* Impossible written consent
* Judiciary protected people
* Minor
* Women of childbearing age without contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Radiation exposure | Immediately post procedure
  Dose area product (cGy/cm2)

SECONDARY OUTCOMES:
Contrast product | Immediately post procedure
  Contrast volume (mL) used during procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No